CLINICAL TRIAL: NCT01930058
Title: A Multiple Dose Study to Evaluate Safety, Pharmacokinetics and Pharmacodynamics of MK-8876 in Hepatitis C Patients
Brief Title: Safety, Pharmacokinetics, and Pharmacodynamics of MK-8876 in Participants With Hepatitis C Infection (MK-8876-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8876-003; 2013-002566-39 (EudraCT Number)
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Panel A: HCV GT3 MK-8876 150 mg (Experimental): Participants infected with HCV GT3 received 150 mg MK-8876 once daily (q.d.) by mouth for 7 days.
  Interventions: Drug: MK-8876
- Panel B: HCV GT3 MK-8876 800 mg (Experimental): Participants infected with HCV GT3 received 800 mg MK-8876 q.d. by mouth for 7 days.
  Interventions: Drug: MK-8876
- Panel E: HCV GT1a MK-8876 800 mg (Experimental): Participants infected with HCV GT1a received 800 mg MK-8876 q.d. by mouth for 7 days.
  Interventions: Drug: MK-8876

INTERVENTIONS:
Drug: MK-8876 — MK-8876 10 mg or 100 mg tablets taken q.d. by mouth.

SUMMARY:
This adaptive design study will evaluate the safety, pharmacokinetics, and effect on hepatitis C virus (HCV) RNA levels of multiple doses of MK-8876 in participants with HCV infection. The study will consist of 4 parts evaluating participants infected with specific hepatitis C virus genotypes and up to 10 panels allowing for additional participants to enroll in each panel as specified in the study analysis. The hypothesis evaluated in the study is that a ≥2.5 log IU/mL reduction in HCV RNA from Baseline will accompany multiple dose administration of MK-8876 in participants with HCV infection.

ELIGIBILITY:
Inclusion Criteria:

* is male, or female of non-childbearing potential (non-childbearing potential is defined as postmenopausal without menses for ≥1 year or after medically documented hysterectomy, oophorectomy, or tubal ligation)
* agrees to use a medically acceptable method of contraception through 90 days after the last dose of study drug if participant has a female partner of childbearing potential must (males should use a condom and their partner of childbearing potential must use hormonal contraception, intrauterine device, diaphragm, cervical cap, or female condom)
* has a body mass index (BMI) between 18 and 37 kg/m^2
* has a clinical diagnosis of chronic HCV infection defined by positive serology for HCV for ≥6 months
* agrees to follow the smoking and other trial restrictions

Exclusion Criteria:

* is mentally or legally institutionalized or incapacitated, has significant emotional problems at study start or has clinically significant psychiatric disorder of the last 5 years
* has a history of clinically significant endocrine, gastrointestinal (except HCV infection), cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* has a history of stroke, chronic seizures, or major neurological disorder
* has a history of cancer (except adequately treated non-melanomatous skin carcinoma, carcinoma in situ of the cervix, or other malignancies which have been successfully treated for ≥10 years
* has a history of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to drugs or food
* has a history of clinically significant hepatic disease, Gilbert's disease, biliary tract disease, or human immunodeficiency virus
* has had major surgery or donated or lost >1 unit of blood within 4 weeks before the study
* has participated in another investigational trial within 4 weeks before the study
* Is unable to refrain from or anticipates the use of any medication from 2 weeks before the study and throughout the study
* consumes >2 glasses of alcoholic beverages per day
* consumes >6 servings (1 serving is ~120 mg caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day
* is a regular user of any illicit drugs or history of drug abuse within 12 months of the study
* has evidence or history of chronic hepatitis not caused by HCV (except acute non-HCV-related hepatitis that resolved >6 months before the study)
* has previously received treatment with another HCV non-nucleoside inhibitor (previous use of other HCV investigational therapies or marketed compounds is permitted if treatment ended ≥3 months before the study)
* has clinical or laboratory evidence of advanced or decompensated liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-10-02 (Actual); Primary Completion 2014-05-05 (Actual); Study Completion 2014-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=8876-003&kw=8876-003

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Panel A: HCV GT3 MK-8876 150 mg | Panel B: HCV GT3 MK-8876 800 mg | Panel E: HCV GT1a MK-8876 800 mg
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Panel A: HCV GT3 MK-8876 150 mg: Participants infected with HCV GT3 received 150 mg MK-8876 q.d. by mouth for 7 days.
- Total: Total of all reporting groups
Arm/Group | Panel A: HCV GT3 MK-8876 150 mg | Panel B: HCV GT3 MK-8876 800 mg | Panel E: HCV GT1a MK-8876 800 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32 (2.6) | 45 (12.5) | 49.7 (7.4) | 42.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in HCV Viral Load
Description: The mean change (log10) in HCV ribonucleic acid (RNA) from baseline to Day 7 was determined for each panel of participants.
Time Frame: Baseline and Day 7
Population: All participants in Panels A, B, and E are included in the analysis.
Measure: Mean (Standard Error); unit: Log10 change
Arm/Group | Panel A: HCV GT3 MK-8876 150 mg | Panel B: HCV GT3 MK-8876 800 mg | Panel E: HCV GT1a MK-8876 800 mg
Number analyzed (Participants) | 3 | 3 | 3
Log10 change | -0.42 (0.12) | -1.88 (0.5) | -3.39 (0.27)

2. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (hr) Post-dose (AUC0-24 hr) of MK-8876
Description: AUC0-24hr is a measure of the mean concentration of drug in plasma after dosing to 24 hr post-dose. Plasma AUC0-24hr was calculated on Day 1 and Day 7 of MK-8876 dosing.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post-dose on Days 1 and 7
Population: All participants in Panels A, B, and E are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM*hr
Arm/Group | Panel A: HCV GT3 MK-8876 150 mg | Panel B: HCV GT3 MK-8876 800 mg | Panel E: HCV GT1a MK-8876 800 mg
Number analyzed (Participants) | 3 | 3 | 3
µM*hr
  Day 1 | 1.9 (88.6) | 4.83 (26.1) | 10.7 (16.5)
  Day 7 | 5.23 (113.7) | 23.1 (13.2) | 23.1 (22.0)

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MK-8876
Description: Cmax is a measure of the maximum plasma concentration of drug post-dose. Plasma Cmax was determined on Day 1 and Day 7 of MK-8876 dosing.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post-dose on Days 1 and 7
Population: All participants in Panels A, B, and E are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Panel A: HCV GT3 MK-8876 150 mg | Panel B: HCV GT3 MK-8876 800 mg | Panel E: HCV GT1a MK-8876 800 mg
Number analyzed (Participants) | 3 | 3 | 3
nM
  Day 1 | 177 (69.7) | 373 (29.7) | 773 (26.1)
  Day 7 | 375 (70.7) | 1310 (12.3) | 1380 (22.9)

4. Secondary Outcome: Trough Plasma Concentration (C24hr) of MK-8876
Description: C24hr is a measure of the plasma drug concentration 24 hours post-dose (i.e., trough concentration). Plasma C24hr was determined on Day 1 and Day 7 of MK-8876 dosing.
Time Frame: 24 hours post-dose on Days 1 and 7
Population: All participants in Panels A, B, and E are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Panel A: HCV GT3 MK-8876 150 mg | Panel B: HCV GT3 MK-8876 800 mg | Panel E: HCV GT1a MK-8876 800 mg
Number analyzed (Participants) | 3 | 3 | 3
nM
  Day 1 | 59.1 (99.5) | 189 (17.1) | 370 (18.2)
  Day 7 | 173 (140.7) | 907 (17) | 869 (21.4)

5. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of MK-8876
Description: Tmax is a measure of time required to reach the maximum plasma drug concentration post-dose. Plasma Tmax was calculated on Day 1 and Day 7 of MK-8876 dosing.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post-dose on Days 1 and 7
Population: All participants in Panels A, B, and E are included in the analysis.
Measure: Median (Full Range); unit: Hours
Arm/Group | Panel A: HCV GT3 MK-8876 150 mg | Panel B: HCV GT3 MK-8876 800 mg | Panel E: HCV GT1a MK-8876 800 mg
Number analyzed (Participants) | 3 | 3 | 3
Hours
  Day 1 | 4 [4 to 6] | 6 [4 to 6] | 4 [4 to 8]
  Day 7 | 4 [4 to 6] | 4 [2 to 6] | 4 [2 to 4]

6. Secondary Outcome: Apparent Terminal Plasma Half-life (t½) of MK-8876
Description: t½ is the time required for the maximum plasma drug concentration to reduce by 50% post-dose. Plasma t½ was determined on Day 7 of MK-8876 dosing.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post-dose on Day 7
Population: All participants in Panels A, B, and E are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Panel A: HCV GT3 MK-8876 150 mg | Panel B: HCV GT3 MK-8876 800 mg | Panel E: HCV GT1a MK-8876 800 mg
Number analyzed (Participants) | 3 | 3 | 3
Hours | 77.1 (20.5) | 140 (24.2) | 62.5 (66.1)

ADVERSE EVENTS:
Time Frame: Up to Day 21
Description: All AE data for GT1a and GT3 participants treated with MK-8876 800 mg were combined.
Groups:
- MK-8876 150 mg: All HCV GT3 participants treated with MK-8876 150 mg are included.
- MK-8876 800 mg: All HCV GT1a and GT3 participants treated with MK-8876 800 mg are included.
Arm/Group | MK-8876 150 mg | MK-8876 800 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 1/3 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8876 150 mg (N=3) | MK-8876 800 mg (N=6)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.